CLINICAL TRIAL: NCT01431118
Title: Iron Metabolism in Dragon Boat Athletes - An Analysis of Changes in Blood Count Parameters Under Sport-specific Stress
Brief Title: Iron Metabolism in Dragon Boat Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: MVZ für Laboratoriumsmedizin Koblenz (Unknown); Deutscher Drachenboot Verband e.V. (Unknown)
Responsible Party: Principal Investigator, Andree Hillebrecht, Dr.med., University of Giessen
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Gi-02-2011
Record Dates: First submitted 2011-08-31; First posted 2011-09-09 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Anaemia
Keywords: iron metabolism; hepcidin; dragon boating; sport-specific stress; iron; anaemia; sport
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sports intervention male (Active Comparator): male athletes of the german national dragon boat team
  Interventions: Other: specific dragon boating training intervention
- sports intervention women (Active Comparator): women athletes of the german national dragon boat team
  Interventions: Other: specific dragon boat intervention

INTERVENTIONS:
Other: specific dragon boating training intervention — male athletes of the german national dragon boat team performing three specific training units at one day
  Arms: sports intervention male
Other: specific dragon boat intervention — women athletes of the german national dragon boat team performing two specific training units and one weight lifting test at one day
  Arms: sports intervention women

SUMMARY:
The purpose of the study is:

* To investigate the effect of sport-specific stress in the iron metabolism of dragon boat athletes
* To investigate the effects of sport-specific stress in the activity of pro-hepcidin and hepcidin

DETAILED DESCRIPTION:
This investigation evaluates the effects of sport-specific stress in iron metabolism of dragon boat athletes. Recent studies showed a significant increase in hepcidin activity under exercise (Röcker L. et al.(2005): Iron regulatory protein hepcidin is increased in female athletes after a marathon. European Journal of Applied Physiology, S. 95, 569-571)which possibly influences the iron metabolism.

In particular in this investigation the activity of pro-hepcidin and hepcidin under sport-specific stress is analysed. Therefore elite dragonboat athletes will be included to this study. Every athlete is tested once. At one exercise day from every athlete the iron metabolism especially the change of hepcidin, prohepcidin and iron before and after a specific dragonboat intervention is analysed.

ELIGIBILITY:
Inclusion Criteria:

* athletes performing dragon boat sport

Exclusion Criteria:

* acute clinically significant intercurrent diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change from Baseline in prohepcidin after performing dragonboating | pre and post exercise intervention at the same day
  one meassurement of prohepcidin immediate before and within three hours after performing two to four specific dragonboat interventions at the same day

SECONDARY OUTCOMES:
haematocrit | pre and post exercise intervention at the same day
  one meassurement of haematocrit immediate before and within three hours after performing two to four specific dragonboat intervention at the same day
value of reticulocytes | pre exercise
  one meassurement of reticulocytes immediate before performing two to four specific dragonboat interventions
value of hypochromic erythrocytes | pre exercise
  one meassurement of hypochromic erythrocytes immediate before performing two to four specific dragonboat interventions
change from Baseline in serum iron after performing dragonboating | pre and post exercise intervention at the same day
  one meassurement of serum iron immediate before and within three hours after performing two to four specific dragonboat interventions at the same day
value of transferrin | pre exercise
  one meassurement of transferrin immediate before performing two to four specific dragonboat interventions
value of transferrin saturation | pre exercise
  one meassurement of transferrin saturation immediate before performing two to four specific dragonboat interventions
value of ferritin | pre exercise
  one meassurement of ferritin immediate before performing two to four specific dragonboat interventions
change from Baseline in hepcidin after performing dragonboating | pre and post exercise intervention at the same day
  one meassurement of hepcidin immediate before and within three hours after performing two to four specific dragonboat interventions at the same day

CONTACTS AND LOCATIONS:
Overall Officials: Andree Hillebrecht, Dr. med., Principal Investigator — Department of sportsmedicine- University Giessen